CLINICAL TRIAL: NCT04943237
Title: Anti-TNF Therapy and Nerve Conduction Studies in Patients With Ankylosing Spondylitis
Brief Title: Anti-TNF Therapy and Nerve Conduction Studies in Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPMRTRHatncsias
Record Dates: First submitted 2021-06-19; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Anti - TNF Therapy; Ankylosing Spondylitis; Neuropathy
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anti-TNF agents — Group of patients using anti-TNF for the last 5 years.
  Other Names: Anti-TNF agents users for the last 5 years.
Drug: Conventional therapy users for the last 5 years — Group of patients not using anti-TNF. Group of patients using conventional therapy (non -steroid anti-inflammatory drugs and/or salazopyrin) for the last 5 years
  Other Names: Conventional therapy (non steroid anti inflammatory drugs and/or salazopyrin)

SUMMARY:
Patients with ankylosing spondylitis were divided into 2 groups as anti-TNF and conventional therapy according to the treatments they were using for the last 5 years. Nerve conduction studies in the upper and lower extremities of the patients were compared.

DETAILED DESCRIPTION:
Demyelinating lesions in central nervous system after anti-TNF agents were reported previously. There are limited studies investigating the effects of anti-TNF treatments on the peripheral nervous system. The aim of this study is to investigate whether peripheral nerves are affected due to long-term use of anti-TNF agents.

Patients with a diagnosis of ankylosing spondylitis who received conventional or anti-TNF therapy for five years at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital were included in the study. The patients were divided into two groups as conventional group and anti-TNF group according to the treatment they received. All patients were evaluated in a single section. Sociodemographic characteristics of the patients and Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functionality Index (BASFI) and Bath Ankylosing Spondylitis Metrology Index (BASMI) scores were recorded. Median-ulnar motor and sensory conduction studies and tibial-peroneal motor and sural nerve sensory conduction studies were performed in both upper extremities of all patients. Median, ulnar, and tibial nerve F-response studies were also performed.

ELIGIBILITY:
Inclusion criteria:

* Patients diagnosed with ankylosing spondylitis
* Patients who have been using conventional therapy (non-steroidal anti-inflammatory drugs and/or salazopyrin) or anti-TNF therapy for more than 5 years.

Exclusion criteria:

* Patients with rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus ......)
* Patients with other systemic diseases that can lead to neuropathy
* Patients who have had a known neuropathy or have taken medication that can lead to neuropathy as a side effect
* Patients with pacemakers

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had the diagnosis of ankylosing spondylitis and had used conventional or anti-TNF therapy at least 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
nerve conduction studies | All patients were evaluated in one session. The assesment of a patient lasted nearly 45-60 minutes
  The evaluation of median, ulnar, tibial, peroneal and sural nerves

CONTACTS AND LOCATIONS:
Overall Officials: Betül Yavuz Keleş, MD, Principal Investigator — Istanbul physical Medicine and Rehabilitation Training and Research Hospital; Ayşe Nur Bardak, prof, Study Director — Istanbul physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and research Hospital, Istanbul, Turkey (Türkiye)